CLINICAL TRIAL: NCT04753502
Title: Laparoscopic Treatment for Appendicitis During Pregnancy: Retrospective Cohort Study
Brief Title: Laparoscopic Treatment for Appendicitis During Pregnancy
Status: Completed | Type: Observational
Sponsor: Austral University, Argentina (Other)
Responsible Party: Principal Investigator, Carina Chwat, Principal Investigator, Austral University, Argentina
Other Study IDs: P20-070
Record Dates: First submitted 2021-02-02; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Other Specified Complications of Pregnancy
Keywords: acute appendicitis; pregnancy; complications
MeSH Terms: conditions — Appendicitis | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laparoscopy — laparoscopic removal of pathologic appendix

SUMMARY:
Acute appendicitis is the most frequent non-obstetric surgical emergency during pregnancy. The benefits of laparoscopy during pregnancy are well known, but complications can occur, and these can affect both the mother and/or the foetus.

Objective: Evaluate results of laparoscopic surgical treatment of acute appendicitis in pregnant women, to analyse the occurrence of adverse postoperative, obstetric and foetal outcomes Methods: Retrospective cohort single-centred observational study on pregnant women with a preoperative diagnosis of acute appendicitis,using computerized medical records' information of pregnant patients admitted to our institution between September 2005 and July 2020

DETAILED DESCRIPTION:
Construction and analysis of the database and study protocol were authorized by the Institutional Evaluation Committee under N° B20-010 and P20-070, respectively.

Assuming a 3: 1 relationship between surgery within 48 hours of symptom onset and surgery after 48 hours of 3: 1, we have an 80% power to find a difference in postoperative morbidity between groups of 30% with error type I of .05.

Analysed variables include: demographic characteristics, gestational age, clinical presentation, symptom duration from onset until surgical resolution, complementary studies, ASA score (Classification of the American Society of Anaesthesiology), intraoperative findings, type of surgery performed, intra and postoperative complications, length of stay, readmissions, use of tocolytics, preterm delivery, birth weight, Apgar score, maternal and foetal mortality, and obstetric and perinatological complications in pregnant patients with a preoperative diagnosis of acute appendicitis.

Any surgery in which the exploratory laparoscopy did not reveal intra-abdominal pathology and the appendix was macroscopically and microscopically normal was classified as a "negative laparoscopy". An "intraoperative complication" was defined as any unexpected intraoperative event, excluding conversion to conventional surgery, which was analysed as an independent event. A "postoperative complication" was defined as any deviation from the usual postoperative course within 30 days of surgery. An "obstetric complication" was one that occurred from the appendectomy until the end of the pregnancy, including foetal death and excluding preterm delivery. Spontaneous abortion and foetal demise were included within the same "foetal loss" outcome. "Preterm labour" was considered to be deliveries or caesarean sections that occurred prior to the 37th week of gestation.

For continuous variables, mean, standard deviation and / or minimum and maximum, or median and interquartile interval (IQR) were used, according to distribution. For categorical variables the number and corresponding percentages were reported. Continuous parameter comparisons were made using the test for independent samples or Wilcoxon-rank test; and when there were more than two groups, Anova or Kruskal Wallis were applied. For the comparison of categorical variables, Chi-square or Fisher's exact test were used, as appropriate. A p <0.05 was considered statistically significant. Likewise, a multivariate analysis was performed for the presence of postoperative and obstetric complications, contemplating possible confounders.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women 18 years or above
* preoperative diagnosis of acute appendicitis
* Diagnosed, operated and followed in Austral University Hospital
* Signed informed consent for surgery and inclusion in databases for further research

Exclusion Criteria:

- Patients operated in another hospital and sent to our institution for postoperative controls.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — participants were pregnant women
Study Population: Pregnant patients of 18 or more years of age admitted to our institution between September 2005 and July 2020 with diagnosis of acute appendicitis.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2005-09-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Postoperative complication | within 30 days of surgery
  Number of participants that present any deviation from the usual postoperative course within 30 days of surgery

SECONDARY OUTCOMES:
obstetric complication | since the appendectomy until date of pregancy termination by vaginal delivery, cesarean section, or foetal death, assesed up to July 2020
  Number of participants that present an obstetric complication from the appendectomy until the end of the pregnancy, including foetal death and excluding preterm delivery

OTHER OUTCOMES:
negative laparoscopy | during laparoscopic abdominal exploration
  Number of participants whose exploratory laparoscopy did not reveal intra-abdominal pathology and the appendix was macroscopically and microscopically normal
foetal loss | since the appendectomy until date of pregancy termination by vaginal delivery, cesarean section, or foetal death, assesed up to July 2020
  Number of participants that present spontaneous abortion or foetal demise
Preterm labour | until 37th week of gestation
  Number of participants with deliveries or caesarean sections that occurred prior to the 37th week of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Carina M Chwat, MD, Principal Investigator — Austral University Hospital
Locations (1):
- Austral University Hospital, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT04753502/Prot_SAP_000.pdf